CLINICAL TRIAL: NCT05862389
Title: Study on the Mechanism of Eating Disorder
Status: Recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1-19-3
Record Dates: First submitted 2023-04-23; First posted 2023-05-17 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
Keywords: Eating disorder; anorexia nervosa; bulimia nervosa; functional magnetic resonance imaging; EEG
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Anorexia nervosa: Patients with anorexia nervosa.
- Bulimia nervosa: Patients with bulimia nervosa.
- Healthy control: The healthy control group

SUMMARY:
Eating disorders (EDs) are severe chronic psychiatric disorders with a not fully understood etiopathogenesis. Previous studies have revealed some biological mechanisms of EDs. However, the etiology and maintenance mechanism of EDs, especially the neuro-mechanisms is still unknown. To explore the pathogenic mechanism and treatment biomarkers of EDs, we design this study. the multidimensional data including the clinicopathological features, neuroimaging data (functional and structural magnetic resonance imaging), electroencephalogram and inflammatory cytokines will be used to investigate the biomarkers for diagnosis and treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

Anorexia nervosa

1. Anorexia nervosa according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5);
2. Age: 13-35 (including 13 and 35)
3. BMI: 13-17.5kg/m^2
4. The participants and/or their legal guardians ( for participants who are younger than 18-year-old) sign the informed consent form voluntarily and agree to participate in all visits and examinations as required by the trial protocol.
5. Do not take any psychiatric medications in past one month.

Bulimia nervosa

1. Bulimia nervosa according to Diagnostic and Statistical Manual of Mental Disorders (5th edition) (DSM-5);
2. Age: 13-35 years old (including 13 and 35)
3. The participants and/or their legal guardians ( for participants who are younger than 18-year-old) sign the informed consent form voluntarily and agree to participate in all visits and examinations as required by the trial protocol.
4. Do not take any psychiatric medications in past one month.

Exclusion Criteria:

1. Patients who meet DSM-5 diagnostic criteria for other mental disorders: Major depressive disorder, anxiety, obsessive-compulsive disorder, personality disorder, mental retardation; drug and/or alcohol dependence;
2. Patients who receive repetitive Transcranial Magnetic Stimulation (rTMS) or modified electroconvulsive therapy (MECT) treatment in past six months.
3. Patients with severe suicidal tendencies or suicidal behavior
4. Pregnant or lactating women;
5. Patients with MRI contraindications;
6. Patients who are regarded as unsuitable by investigators for this clinical trial.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients who are diagnosed with anorexia nervosa and bulimia nervosa.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The change of severity of illness at 8 weeks | Day 0 to Day 56
  The change of scores of Eating disorder Inventory (EDI) will be used to estimate the change of severity of illness. The scores of 8-week will be compared with those of baseline. The maximum of EDI is 396 and the minimum score is 0.
The change of eating disorder behaviors and cognition | Day 0 to Day 56
  The change of scores of Eating Disorder Examination Questionnaire (EDEQ) will be used to estimate the change of behaviors and cognition during treatment.The maximum score of EDEQ is 32.5 and the minium score is 0.

SECONDARY OUTCOMES:
The change of severity of illness at early or later timepoints during treatment | Day 0 to Day 28; Day 0 to Month 3; Day 0 to Month 6; Day 0 to Month 12
  The change of scores of Eating disorder Inventory (EDI) will be used to estimate the change of severity of illness. The maximum of EDI is 396 and the minimum score is 0
The change of eating disorder behaviors and cognition | Day 0 to Day 28; Day 0 to Month 3; Day 0 to Month 6; Day 0 to Month 12
  The change of scores of Eating Disorder Examination Questionnaire (EDEQ) will be used to estimate the change of behaviors and cognition during treatment.The maximum score of EDEQ is 32.5 and the minium score is 0.

CONTACTS AND LOCATIONS:
Overall Officials: Tian-Mei Si, Ph.D, Study Director — Peking University Sixth Hospital
Locations (1):
- Institute of Mental Health, Peking University Sixth Hospital, Beijing, China